CLINICAL TRIAL: NCT04341987
Title: Treating Nightmares Among Veterans Health Administration Domiciliary Patients
Brief Title: Treating Nightmares Among Domiciliary Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-related
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1534869
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Nightmare
Keywords: nightmares; treatment; substance use; imagery rehearsal therapy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brief Imagery Rehearsal Therapy (Experimental): The brief two-session, behaviorally-based imagery rehearsal intervention is based on components from previous group and individual formats that have been published, but will be presented in an abbreviated manner. In the first session, Veterans will be presented with psychoeducation about dreaming, basics of sleep hygiene and stimulus control techniques, how to change negative dreams from a "learned habit" perspective, re-scripting, and how to rehearse new dream imagery. They will then be asked to complete in-session practice of imagery rehearsal with the new imagery developed. Veteran will be instructed in practice post-session.
  Interventions: Behavioral: brief Imagery Rehearsal Therapy
- Treatment As Usual (Other): Patients in this condition are free to receive treatment as usual for nightmares, which may be a medication, supportive counseling or no treatment.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: brief Imagery Rehearsal Therapy — Two-sessions of behaviorally-based imagery rehearsal therapy.
  Arms: brief Imagery Rehearsal Therapy
Other: Treatment As Usual — may include medication treatment or behavioral treatment for nightmares other than imagery rehearsal therapy
  Arms: Treatment As Usual

SUMMARY:
The purpose of the study is to assess the efficacy of a 2-session intervention to reduce nightmares among Veterans admitted VA mental health residential rehabilitation treatment programs.

DETAILED DESCRIPTION:
Sleep disturbances and suicide are highly prevalent among Veterans and recent research also suggests high comorbid rates of sleep and suicide in Veterans discharged from VA mental health residential rehabilitation treatment programs (MHRRTP; domiciliaries). Nightmares are a frequent concern identified by MHRRTP patients and are a modifiable risk factor for suicide risk. Little is known, however, about the treatment of nightmares and subsequent impact in this setting. The primary aims of the present project are to investigate the efficacy and acceptability of delivering a 2-session intervention to reduce nightmares among Veterans admitted to a MHRRTP. This study will examine this intervention's impact on reducing nightmare distress and nightmare frequency, as well as assess treatment acceptability. Changes in suicide risk following intervention will also be explored. This research will be conducted within the Canandaigua and Bath VA domiciliary programs which currently accommodate ~150-175 Veterans. The study will be a randomized control trial with a hybrid design that uses stratification based on prescription use and randomly assigns individuals (N = 48) to either the treatment group or treatment as usual group (TAU). Veterans referred for the protocol will be screened for eligibility and then if appropriate, scheduled for a baseline evaluation, randomized to either the treatment group or TAU group, seen for two intervention sessions one week apart, and then be followed up with 4- and 8-weeks post initial treatment via telephone. This research has potential to highlight valuable targets for cross-cutting treatment in a rehabilitation setting that can be delivered in civilian and Veteran samples.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* endorses nightmares at least once a week
* score of 10 or greater on the Disturbing Dreams and Nightmares Severity Index

Exclusion Criteria:

* unable to consent
* diagnosis of serious mental illness (schizophrenia, schizoaffective disorder)
* active suicide ideation with plan and intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Nightmare Frequency | Change in total nights with nigthmares in the past week from baseline to 8 week follow-up.
  Disturbing Dreams and Nightmares Severity Index. The score for frequency ranges from 0-7.
Nightmare Severity | Change in nigthmare severity from baseline to 8 week follow-up.
  Disturbing Dreams and Nightmares Severity Index. The score for severity ranges from 0-6.

CONTACTS AND LOCATIONS:
Overall Officials: WIlfred R Pigeon, PhD, Principal Investigator — Canandaigua VAMC

IPD SHARING:
Plan to Share IPD: No
Because the potential participant pool is relatively small (inpatients in a specific location during a specific time period) individuals are potentially identifiable even if data are de-identified.